CLINICAL TRIAL: NCT00990444
Title: A Double-Blind Two Part Placebo-Controlled Study Consisting of a Single Ascending and Multiple-Dose Tolerance Study of Peroral Insulin in Patients With Type 2 Diabetes
Brief Title: A Two Part Study of Peroral Insulin in Type 2 Diabetes
Acronym: ORA2
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bows Pharmaceuticals AG (Industry)
Responsible Party: Nabil Al-Tawil, Karolinska Trial Alliance
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORA2-2009-010660-42
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-10

CONDITIONS: Diabetes Mellitus
Keywords: blood glucose; blood insulin; dextran; diabetes; hyperglycemia; hypoglycemia; oral delivery; portal delivery
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia; Hypoglycemia | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Treatment with vehicle capsule containing excipients only, taken in conjunction with standard meal.
  Interventions: Drug: Insulin in Dextran Matrix
- Oral Insulin in Dextran (Active Comparator): Treatment with fixed insulin dose taken in conjunction with standard meal.
  Interventions: Drug: Insulin in Dextran Matrix

INTERVENTIONS:
Drug: Insulin in Dextran Matrix — Fixed dose capsule with 100 IU of insulin in dextran matrix. Investigational drug or placebo are administered in conjunction with food intake on a background of metformin.
  Other Names: Peroral insulin

SUMMARY:
Insulin is normally not bioavailable when taken through the oral route, as degradation of the molecule may occur both in the ventricle and in the intestine. Oral administration with uptake from the lesser intestine would offer major advantages if made possible. It would offer a simple non-injection method to administer insulin in connection with a meal and absorbed insulin would enter the blood stream and mimic the natural distribution in the body with a first pass through the liver. The sponsor of this study has developed a novel oral insulin formulation that is based on a proprietary dextran matrix. The investigational drug is a capsule containing 100 IU of human insulin in dextran matrix.

The primary objective of this study is to establish the safety, tolerance and PD profile (i.e. pharmacodynamic parameters for glucose and insulin) of peroral insulin in dextran matrix in patients with type 2 diabetes.

The phase I/II study protocol consists of two parts; part 1 (dose finding) and part 2 (dose verification). In study part 1 single escalating doses of oral insulin or placebo is given to the test subjects. Capillary blood glucose is used to assess the insulin effect. Subsequently, in study part 2, the investigational drug will be administered 3 times daily on 6 consecutive days. The starting dose of part 2 will be the lowest effective dose found in study part 1. Dose escalation will be done in increments of 100 IU. The total number of subjects will be 32 (for part 1 and 2 combined).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with Type 2 diabetes who were diagnosed for a minimum of 6 months, age 30-65 years.
* Subjects on a stable dose of metformin for at least two months with a total daily dose of

  ≤ 2600 mg/day.
* Subjects demonstrating an insulin resistance value (IR) lower than 3 based on the HOMA-2 model (University of Oxford, 2004) at Screening 2.
* Hemoglobin A1c <9%.
* Fasting capillary blood glucose within the range 6.0-9.0 mmol/L (108-162 mg/dL) at Screening 1, Screening 2 and Randomization visit. For study Part 1 only, the maximum and minimum of these three measurements may not differ by more than 2 mmol/L.
* Body Mass Index (BMI) of 25-32 kg/m2
* Medically stable as determined by history and physical examination, including vital signs.
* Screening laboratory tests must be within normal range or judged as not clinically significant by Principal investigator/Subinvestigator.
* Negative urine ketoacidosis test
* ECG including QTcB shows no clinically significant abnormality or acute ischemia
* Supine BP ≤ 160/100 mm Hg diastolic/systolic.
* Able to adhere to the study visit schedule, and to understand and comply with other protocol requirements.
* Capable of giving informed consent, which must be obtained prior to any screening procedures.
* Non user of tobacco products for a minimum of 6 months prior to the first dose.
* Negative urine screen for drugs of abuse and an alcohol breath test at screening and check in.
* Negative laboratory screen for Hepatitis B (HBsAg and anti-HBc antibodies), Hepatitis C (anti HCV) and HIV (1&2).
* Not on any prohibited medication, including alcohol.
* Female subjects willing to use adequate method of contraception from the time of the first dose until one month after the last dose.
* Willing to eat standard meal in accordance with the protocol.

Exclusion Criteria:

* History of significant coronary disease or renal failure
* Other significant medical problems that would preclude participation in a clinical trial
* Participation in a clinical trial within the prior 3 months
* History of GI surgery or known GI motility disorders.
* History of a serious infection, including but not limited to hepatitis, pneumonia, or pyelonephritis, or have been hospitalized or received intravenous antibiotics for an infection, during the previous two months.
* A chronic or recurrent infectious disease, including but not limited to, chronic renal infection, chronic chest infection (bronchiectasis), sinusitis, recurrent urinary tract infection (recurrent pyelonephritis or chronic nonremitting cystitis), open skin wound, or ulcer.
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine (other than diabetes), pulmonary, cardiac, neurologic, or cerebral disease, or any other condition which increases risk of participation in this trial in the opinion of the investigator.
* Currently known malignancy or a history of malignancy within the previous 5 years.
* History of polyps in the gastrointestinal tract.
* Known to have had a substance abuse (drug or alcohol) problem within the previous 5 years
* Unable to undergo venipunctures for study purposes because of poor tolerability or lack of easy access.
* Engaging in any strenuous exercise (such as running or weight lifting or playing any team sports such as soccer for 48 hours prior to admission to the inpatient unit and no strenuous exercise will be permitted for the duration of the study (applies to both part 1 and part 2).
* Donation or loss of 400 ml blood or more within 3 months prior to the first dose or donation of plasma within 7 days prior to the first dose.
* Difficulty in swallowing capsules.
* A recent adult history of clinically significant allergic reaction to any drug.
* Any other medical condition that, in the opinion of the investigator, disqualifies the subject.
* Female subject with positive pregnancy test at screening, Day -1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Identification of the lowest dose of oral insulin in dextran matrix that produces a significant lowering of post-prandial blood glucose. | 6 hours

SECONDARY OUTCOMES:
To establish the dose(s) when administered in a multi-dose fashion that lowers plasma glucose levels versus placebo in patients with Type 2 diabetes | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Al-Tawil, M.D.; Ph.D., Principal Investigator — Karolinska Trial Alliance
Locations (1):
- Karolinska Trial Alliance, Phase I Unit, Stockholm, Solna, Stockholm, Sweden